CLINICAL TRIAL: NCT03336242
Title: A Phase 2, Open-label, Dose-finding Study to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of Pharmaceutical Grade Synthetic Cannabidiol Oral Solution in Pediatric Patients With Treatment-Resistant Childhood Absence Seizures
Brief Title: Cannabidiol Oral Solution in Pediatric Participants With Treatment-Resistant Childhood Absence Seizures
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: More patients in Cohort 1 than Cohort 2 demonstrated a clinically meaningful reduction of seizure count. Given this, enrollment of Cohort 3 was discontinued.
Sponsor: Radius Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INS011-17-103
Record Dates: First submitted 2017-10-31; First posted 2017-11-08 (Actual); Results first posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Childhood Absence Epilepsy
MeSH Terms: conditions — Epilepsy, Absence | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Cannabidiol Oral Solution 20 mg/kg/day (Experimental): Treatment Period: Cannabidiol Oral Solution 20 milligrams per kilogram per day (mg/kg/day) divided twice daily (BID) for 4 weeks.
  Interventions: Drug: Cannabidiol Oral Solution
- Cohort 2: Cannabidiol Oral Solution 30 mg/kg/day (Experimental): Titration Period: Cannabidiol Oral Solution 20 mg/kg/day divided BID for 5 days.
  Treatment Period: Cannabidiol Oral Solution 30 mg/kg/day divided BID for 4 weeks.
  Interventions: Drug: Cannabidiol Oral Solution
- Cohort 3: Cannabidiol Oral Solution 10 mg/kg/day (Experimental): Treatment Period: Cannabidiol Oral Solution 10 mg/kg/day divided BID for 4 weeks.
  Interventions: Drug: Cannabidiol Oral Solution

INTERVENTIONS:
Drug: Cannabidiol Oral Solution — An oral solution containing pharmaceutical grade cannabidiol (nonplant-based).

SUMMARY:
The primary purpose of this study is to assess the efficacy of Cannabidiol Oral Solution in the treatment of pediatric participants with treatment-resistant childhood absence seizures. This study will also assess safety, tolerability and pharmacokinetics of Cannabidiol Oral Solution, and any improvement in qualitative assessments of participant status over the duration of the study in pediatric participants with treatment-resistant childhood absence seizures. The study will include a 4-week Screening Period, a 5 or 10 day Titration Period (depending study Cohort), a 4-week Treatment Period followed by 5-day Tapering for doses >20 mg/kg/day and a 4-week Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

1. Patient and/or parent(s)/caregiver(s) fully comprehend the informed consent form and assent form, understand all study procedures, and can communicate satisfactorily with the investigator and study coordinator, in accordance with applicable laws, regulations, and local requirements.
2. Male or female between 3 and 12 years (inclusive) at the time of onset and between 3 and 17 years of age (inclusive) at the time of consent.
3. Body weight ≥ 10 kg.
4. Diagnosed with childhood absence epilepsy, confirmed by electroencephalogram (EEG) with at least 3 bursts of general spike wave of 2.7 to 5 hertz lasting ≥3 seconds during the 4-hour EEG, and has had an adequate trial of at least 2 antiepileptic drugs (AEDs) and are treatment-resistant to at least one AED.
5. Willingness to not start a ketogenic diet during the Baseline or Treatment Period.
6. A female patient is eligible to participate in the study if she is premenarchal, or of childbearing potential with a negative urine pregnancy test at the Screening Visit. If sexually active, she must agree to either complete abstinence from intercourse or use acceptable methods of contraception throughout the study and for 4 weeks after completion of study participation or discontinuation from investigational product.
7. A sexually active male patient must be willing to use acceptable methods of contraception throughout the study and for 4 weeks after completion of study participation or discontinuation from investigational product.
8. In the opinion of the investigator, the parent(s)/caregiver(s) is willing and able to comply with the study procedures and visit schedules and the Follow-up Visits.
9. General good health based on physical and neurological examinations, medical history, and clinical laboratory values completed during the Screening Visit that would prohibit the patient from safely participating in the trial as judged by the investigator.

Exclusion Criteria:

1. Patient or parent(s)/caregiver(s) have daily commitments during the study duration that would interfere with attending all study visits.
2. Has a history of nonfebrile seizures other than absence seizures.
3. Has a history of febrile seizures after 3 years of age.
4. Has a history consistent with juvenile absence epilepsy or juvenile myoclonic epilepsy.
5. Currently taking felbamate.
6. Currently taking phenytoin, fluvoxamine, carbamazepine, or St. John's Wort.
7. Currently taking concomitant medications that are strong inhibitors/inducers/sensitive substrates with a narrow therapeutic index for cytochrome P450 3A4 (CYP3A4), CYP2C9, or CYP2C19. (Stable doses of Valproic Acid during the screening, titration, treatment, and follow-up periods are permitted).
8. Currently on a ketogenic diet.
9. In the opinion of the investigator, any clinically significant, unstable medical abnormality, chronic disease, or a history of a clinically significant abnormality of the cardiovascular, gastrointestinal, respiratory, hepatic, or renal systems.
10. Clinically significant abnormal liver function test (LFT) values, including albumin, direct bilirubin, total bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) ≥3 times the upper limit of normal (ULN).
11. History or presence of abnormal electrocardiograms (ECGs) that are clinically significant in the opinion of the investigator.
12. Has a current or history of clinically significant intellectual disability or major psychiatric disease, including autism spectrum disorder, which would interfere with compliance.
13. For patients aged 7 to 17 years of age and for whom the Columbia Suicide Severity Rating Scale (C-SSRS) is developmentally appropriate, an affirmative answer to queries regarding active suicidal ideation with some intent to act but without a specific plan or active suicidal ideation with a specific plan and intent on the C-SSRS assessment at the Screening Visit.
14. Any history of attempted suicide.
15. Previously received any investigational drug or device or investigational therapy within 30 days before Screening.
16. Taken any cannabinoids in the 30 days prior to the Screening Visit.
17. History of an allergic reaction or a known or suspected sensitivity to any substance that is contained in the investigational product formulation.
18. Known infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
19. In the opinion of the investigator, the patient is unsuitable in any other way to participate in this study.
20. Body weight <10 kg or >90 kg.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elkashef, MD, Study Director — INSYS Therapeutics Inc
Locations (11):
- United States (11):
  - Nicklaus Children's Hospital, Miami, Florida
  - Pediatric Epilepsy and Neurology Specialists, Tampa, Florida
  - Clinical Integrative Research Center of Atlanta, Atlanta, Georgia
  - Clinical Research Center of Nevada, Henderson, Nevada
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Akron Children's Hospital, Akron, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Specialty Group, Division of Child & Adolescent Neurology, Norfolk, Virginia
  - Research and Innovation/MultiCare Health System, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Sponsor terminated the study and no participants were enrolled in Cohort 3.
Groups:
- Cohort 1: Treatment Period: Cannabidiol Oral Solution 20 milligrams per kilogram per day (mg/kg/day) divided twice daily (BID) for 4 weeks.
  Cannabidiol Oral Solution: An oral solution containing pharmaceutical grade cannabidiol (nonplant-based).
- Cohort 2: Titration Period: Cannabidiol Oral Solution 20 mg/kg/day divided BID for 5 days.
  Treatment Period: Cannabidiol Oral Solution 30 mg/kg/day divided BID for 4 weeks.
  Cannabidiol Oral Solution: An oral solution containing pharmaceutical grade cannabidiol (nonplant-based).
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled and received at least 1 dose of study drug. No participants enrolled in Cohort 3.
Groups:
- Cohort 1: Treatment Period: Cannabidiol Oral Solution 20 mg/kg/day divided BID for 4 weeks.
  Cannabidiol Oral Solution: An oral solution containing pharmaceutical grade cannabidiol (nonplant-based).
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.8 (2.74) | 8.0 (3.02) | 8.4 (2.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Absence Seizure Counts Assessed by Video-electroencephalogram (EEG) at Visit 5
Description: A 4-hour video-EEG was performed for all participants at Baseline, during the Treatment Period, and at the End of the Study/Early Withdrawal Visit. Hyperventilation was conducted during the video-EEG to count the number of absence seizures. A negative change value indicates an improvement in seizure activity. A positive change value indicates a worsening in seizure activity. Percent change from baseline was calculated as (100*(week 4-baseline)/baseline).
Time Frame: Baseline (Visit 2, Day 1 of Titration Period) and Visit 5 (Week 4, Day 6 of Treatment Period)
Population: The Sponsor terminated this study and no participants were enrolled on Cohort 3.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 10 | 9
percent change | 40.67 (180.919) | 35.12 (121.518)

2. Primary Outcome: Percent Change From Baseline in Time to Absence Seizure During Hyperventilation Testing on Video-EEG at Visit 5
Description: A 4-hour video-EEG was performed for all participants at Baseline, during the Treatment Period, and at the End of the Study/Early Withdrawal Visit. Hyperventilation was conducted during the video-EEG to count the number of absence seizures. Percent change from baseline calculated as (100*(week 4-baseline)/baseline).
Time Frame: Baseline (Visit 2, Day 1 of Titration Period) and Visit 5 (Week 4, Day 6 of Treatment Period)
Population: The Sponsor terminated this study and no participants were enrolled on Cohort 3.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 9 | 8
percent change | 162.24 (344.028) | 64.51 (115.502)

3. Primary Outcome: Number of Participants Seizure-Free at Visit 5
Description: Daily seizure activity was recorded in a diary. Each day, the participant or parent/caregiver responded to the question: "How many absence seizures did the patient have today?".
Time Frame: Visit 5 (Week 4, Day 6 of Treatment Period)
Population: The Sponsor terminated this study and no participants were enrolled on Cohort 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 10 | 9
Participants | 1 | 0

4. Primary Outcome: Clinical Global Impression of Improvement (CGI-I) Score at Visit 5
Description: The CGI-I questionnaire was completed by the parents/caregivers and the investigator and was used to assess participants' global status of their condition at Week 4 of the Treatment Period using a 7-point scale, where 1=very much improved and 7=very much worse since the initiation of treatment.
Time Frame: Visit 5 (Week 4, Day 6 of Treatment Period)
Population: The Sponsor terminated this study and no participants were enrolled on Cohort 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 10 | 10
units on a scale | 2.9 (0.88) | 3.1 (0.99)

5. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a patient administered a pharmaceutical product during the course of a clinical investigation. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product, whether or not thought to be related to the investigational product. A treatment-emergent AE is an AE with onset that occurs after receiving study drug. A SAE is any untoward medical occurrence that results in death, is life-threatening, requires the participant be at a risk of death at the time of the event, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality/birth defect, or other serious event that requires medical or surgical intervention. A summary of SAEs and all other non-serious AEs, regardless of causality, is located in the Reported AEs module.
Time Frame: Day 1 (after dosing) up to Visit 7 (Week 4 of the Follow-Up Period)
Population: All participants who were enrolled and received at least 1 dose of study drug. The Sponsor terminated this study and no participants were enrolled on Cohort 3.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 10 | 10
participants
  Number of participants with AEs | 6 | 7
  Number of participants with SAEs | 0 | 0

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) and Dose-normalized Cmax (Cmax/D) for Cannabidiol Under Fed and Fasted Conditions
Description: The Cmax and Cmax/D for cannabidiol were evaluated under fed and fasted conditions.
  Fed: Participant arrived at the site on Day 1 of Week 4 of the Treatment Period without food and the morning dose. The site provided a high fat/high-calorie food and then dosed the participant. Blood samples were collected pre-dose (before meal/morning dose) and 2, 4, and 6 hours after the morning dose (but before the next dose).
  Fasted (2 hours before dose until 2 hours after dose): Participants arrived at the site on Day 2 of Week 4 of the Treatment Period without food and the morning dose. The site provided a standard meal 2 hours after the dose. Blood samples were collected pre-dose and 2 (before meal), 4, 6 hours after the morning dose (but before the next dose).
Time Frame: Visit 3 (Week 1, Day 1 of Treatment Period; Pre-dose, 2, 4, 6 Hours Post-dose), Visit 5 (Week 4, Day 6 of Treatment Period; Pre-dose, 2, 4, 6 Hours Post-dose), and Visit 6 (Week 4, Day 7 of Treatment Period; Pre-dose, 2, 4, 6 Hours Post-dose)
Population: The Sponsor terminated this study and no participants were enrolled in Cohort 3. No data was collected for any pharmacokinetic analysis, therefore no clinical data will be reported on this outcome measure.
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Area Under the Plasma Concentration Curve From Time 0 to the Last Measured Concentration (AUC(0-t)) and Dose Normalized AUC(0-t) [AUC(0-t)/Dose] for Cannabidiol Under Fed and Fasted Conditions
Description: The AUC(0-t) and AUC(0-t)/dose for cannabidiol were evaluated under fed and fasted conditions.
  Fed: Participant arrived at the site on Day 1 of Week 4 of the Treatment Period without food and the morning dose. The site provided a high fat/high-calorie food and then dosed the participant. Blood samples were collected pre-dose (before meal/morning dose) and 2, 4, and 6 hours after the morning dose (but before the next dose).
  Fasted (2 hours before dose until 2 hours after dose): Participants arrived at the site on Day 2 of Week 4 of the Treatment Period without food and the morning dose. The site provided a standard meal 2 hours after the dose. Blood samples were collected pre-dose and 2 (before meal), 4, 6 hours after the morning dose (but before the next dose).
Time Frame: as for outcome 6
Population: as for outcome 6
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Trough Plasma Concentration (Ctrough) and Dose Normalized Ctrough (Ctrough/Dose) for Cannabidiol Under Fed, Fasted, and Normal Conditions
Description: The Ctrough and Ctrough/dose for cannabidiol were evaluated under fed, fasted, and normal conditions.
  Fed: Participant arrived at the site on Day 1 of Week 4 of the Treatment Period without food and the morning dose. The site provided a high fat/high-calorie food and then dosed the participant. Blood samples were collected pre-dose (before meal/morning dose) and 2, 4, and 6 hours after the morning dose (but before the next dose).
  Fasted (2 hours before dose until 2 hours after dose): Participants arrived at the site on Day 2 of Week 4 of the Treatment Period without food and the morning dose. The site provided a standard meal 2 hours after the dose. Blood samples were collected pre-dose and 2 (before meal), 4, 6 hours after the morning dose (but before the next dose).
Time Frame: as for outcome 6
Population: as for outcome 6
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) up to Visit 7 (Week 4 of the Follow-Up Period
Description: Safety population included all participants who received at least 1 dose of study medication.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 7/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=10) | Cohort 2 (N=10)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (7)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Coordination abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was prematurely terminated by the Sponsor. Enrollment of Cohort 3 was discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT03336242/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT03336242/SAP_001.pdf